CLINICAL TRIAL: NCT03388255
Title: A Phase IV, Single-arm, Open-label Clinical Trial to Evaluate the Efficacy and Safety of PLACENTEX ® Polydeoxyribonucleotide i.m. in Patients With Fibrotic and Atrophic Cutaneous Lesions in Scleroderma Diseases
Brief Title: Efficacy and Safety of PLACENTEX ® i.m. in Patients With Scleroderma Diseases
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: the clinical center has too much difficulty recruiting as a rare condition
Sponsor: Mastelli S.r.l (Industry)
Collaborators: Sintesi Research Srl (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PDRN-01-16
Record Dates: First submitted 2017-12-21; First posted 2018-01-02 (Actual); Last update posted 2021-09-16 (Actual); Status verified 2021-09

CONDITIONS: Scleroderma Disease
Keywords: Polydeoxyribonucletide; Placentex; PDRN
MeSH Terms: conditions — Scleroderma, Diffuse | interventions — Polydeoxyribonucleotides

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Polydeoxyribonucleotides (Experimental): PLACENTEX: Polydeoxyribonucleotides 5.625 mg/3 ml for parenteral use i.m.
  The study period consists of the following phases:
  * Treatment period: 3 months (daily i.m. treatment with PLACENTEX ® Polydeoxyribonucleotide 5.625 mg/3 ml for parenteral use, one vial per day for intra-muscular administration).
  * Follow up period: 3 months after end of active treatment, without study medication.
  Interventions: Drug: Polydeoxyribonucleotides

INTERVENTIONS:
Drug: Polydeoxyribonucleotides — Polydeoxyribonucleotide 5.625 mg/3 ml for parenteral use i.m.
  The study period consists of the following phases:
  * Treatment period: 3 months (daily i.m. treatment with PLACENTEX ® Polydeoxyribonucleotide 5.625 mg/3 ml for parenteral use, one vial per day for intra-muscular administration).
  * Follow up period: 3 months after end of active treatment, without study medication.
  Other Names: PLACENTEX

SUMMARY:
This is a phase IV, single-arm, open-label clinical trial to evaluate the efficacy and safety of PLACENTEX ® Polydeoxyribonucleotide i.m. in patients with fibrotic and atrophic cutaneous lesions in scleroderma diseases during the inactive stage of the disease (experiencing dystrophic outcomes of the disease with no inflammatory component at the time of enrolment).

The patients enrolled will be evaluated at study site at screening (V1), then after 3 months of treatment with PLACENTEX ® Polydeoxyribonucleotide (one vial per day for intra-muscular administration) (V2). After completion of the study treatment period, the patients will be followed for an additional period of 3 months without study medication, after which the patient will visit the site for the last visit (V3). 1 investigational site. 45 patients enrolled (included drop-outs).3 months of treatment with PLACENTEX ® Polydeoxyribonucleotide (one vial per day for intra-muscular administration).

DETAILED DESCRIPTION:
This is a phase IV, single-arm, open-label clinical trial to evaluate the efficacy and safety of PLACENTEX ® Polydeoxyribonucleotide 5.625 mg/3 ml for parenteral use i.m. in patients with fibrotic and atrophic cutaneous lesions in scleroderma diseases during the inactive stage of the disease (experiencing dystrophic outcomes of the disease with no inflammatory component at the time of enrolment). A total of n. 45 patients (including drop-outs, who will not be replaced) will be enrolled in this study.

The patients enrolled will be evaluated at study site at screening (V1), then after 3 months of treatment with PLACENTEX ® Polydeoxyribonucleotide 5.625 mg/3 ml for parenteral use (one vial per day for intra-muscular administration) (V2). After completion of the study treatment period, the patients will be followed for an additional period of 3 months without study medication, in which the patient will visit the site for the last visit (V3).

The IMP units will be dispensed to the patient at the study site at visit 1 (Screening Visit). Patients will be instructed to store IMP at room temperature and to return all used empty secondary packages and unused IMP units at visit 2 (End of Treatment Visit), at this time the Investigator/site coordinator will assess the patient's compliance with the prescribed regimen for the study medication. Compliance with the dosing regimen will be determined by performing IMP accountability of returned boxes of the IMP used and IMP unused units at visit 2 (End of Treatment Visit). Accountability records will be maintained during the study.

In order to prevent any interference in the evaluation of PLACENTEX ® Polydeoxyribonucleotide 5.625 mg/3 ml by prior therapies (corticosteroids, immune-suppressive agents) a wash-out period of 1 month has been planned before starting the investigational treatment. Such period will allow also to be definitely sure of the stability of inactive stage of the disease.

Treatment with steroid therapy and/or systemic immunosuppressive therapy within 1 month prior to screening visit are therefore not allowed. Additionally, the patient will be requested not to take local/systemic corticosteroids or local/systemic immunosuppressive therapy during the study period.

In case of non-response to the treatment with PLACENTEX ® or in case of worsening of the disease, the patient will be withdrawn from the study and an alternative treatment will be considered by Investigator on a case-by-case basis.

During the study period the following assessments will be performed:

* Photography of target cutaneous lesion, to record size and location.
* Tele-thermography of target cutaneous lesion, to record the characteristics of heat loss and store TT images of the lesion.
* Ultrasound evaluation of target cutaneous lesion, to record the subcutaneous measuring parameters indicative of the disease (thickness of subcutaneous adipose layer, etc.)
* Clinical evaluation of patient's cutaneous lesions. A score (LOSCAT Score) from 0 (none) to 3 (high) will be calculated with regard to the presence of atrophy and sclerosis.
* A biopsy sample will be collected from target cutaneous lesion for subsequent histological analysis. A score from 0 (none) to 3 (high) will be calculated with regard to the presence of epidermal, dermal, hypodermic and skin appendages atrophy as well as dermal and hypodermic sclerosis.
* A self-administered Dermatology Life Quality Index (DLQI) from patient, to collect information with particular regard to quality of life, difficulty in walking, loss of function.
* Evaluation of the target cutaneous lesion through a SkinFibrometer, to measure the degree of induration of skin.
* Vital signs will be measured.
* Concomitant medications and medical history will be recorded.

Local laboratory assessments will be performed in order to confirm the safety of the drug treatment, as absence of inflammation or clinical worsening following treatment with drug, according to Investigator's judgment. When abnormal laboratory values or test results constitute an adverse event (i.e., induces clinical signs/symptoms or requires therapy) they must be recorded on the Adverse Events e-CRF page.

Vital signs (heart rate and blood pressure) will be completed at screening visit. Blood pressure and heart rate will be recorded in a sitting position after resting for 5 minutes, instead Physical examination will be performed at all scheduled visits. Significant findings present prior to the start of the study medication treatment must be included in the relevant medical history or current medical history condition in the e-CRF.

Significant findings after the start of the study which meet the definition of an adverse event must be recorded in appropriate place in the e-CRF and evaluated by the Investigators.

In the study, any event occurring after that patient has signed the Informed Consent, should be considered and recorded as an AE. Adverse events, especially those for which the relationship to the study drug is possible, probable or remote, should be followed up until they have stabilized.The Sponsor, via PhV responsabile is responsible for reporting all applicable SAEs and SUSARs to Regulatory authorities, Investigators, and IECs, as applicable, in accordance with national regulations in the countries where the study is conducted.

All analyses will be performed using SAS v. 9.2 (Statistical Analysis System - New Cary USA) or later in Microsoft Windows 7 Professional environment.

For patients with missing values will be applied the Last Observation Carried Forward (LOCF) approach. All variables will be summarized using appropriate descriptive statistics (mean, standard deviation, median and range for continuous variables, and frequencies and percentages for categorical variables) followed by the calculation of 95% Confidence interval, if pertinent and applicable. A two-tailed alpha level of 0.05 will be used for each statistical test. All treated patients will be included in the Intention-To-Treat population (ITT).

ELIGIBILITY:
Inclusion Criteria:

1. Male or female age > 18 years.
2. Patients diagnosed with localized scleroderma diseases during inactive stage with fibrotic and atrophic cutaneous lesions confirmed histologically.
3. Understanding the nature of the study and Signature of the written informed consent.
4. Negative pregnancy test at study entry for females of child bearing potential.
5. If the patient is a female of childbearing potential (less than 24 months since the last menstrual bleeding), she is using an acceptable and effective method of contraception during the study period.

Exclusion Criteria:

1. Patients under treatment with steroid therapy and/or systemic immunosuppressive therapy within 1 month prior to screening.
2. Patients with ongoing infectious processes at the level of target lesions.
3. Women who are pregnant or breast feeding.
4. Know allergy or hypersensitivity to the active principle of the investigational drug or to one of its excipients.
5. Patients with a condition or concurrent severe and/or uncontrolled medical disease which could compromise his/her participation, compliance with and/or completion of study procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2016-11-08 (Actual); Primary Completion 2019-10-30 (Actual); Study Completion 2019-10-31 (Actual)

PRIMARY OUTCOMES:
Localized Scleroderma Cutaneous Assessment Tool - LOSCAT | 6 months
  The LoSCAT assesses 18 cutaneous anatomic sites, capturing both disease activity (mLoSSI) and damage (LoSDI) parameters. This score will take into consideration all the cutaneous lesions resulting from localized scleroderma diseases during the inactive stage of the disease.Scores for each site are based on the most severe score for each parameter. In order to minimize inter-subject variability, all skin changes are compared with the contralateral or ipsilateral skin area.

SECONDARY OUTCOMES:
tele-thermographic profile | 6 months
  Changes in the tele-thermographic profile of target cutaneous lesion following treatment with drug, according to Investigator's judgment
ultrasound profile | 6 months
  Changes in the ultrasound profile of target cutaneous lesion following treatment with drug, according to Investigator's judgment.
histology improvement | 3 months
  Measurement of histology improvement of target cutaneous lesion following treatment with drug through a validated score ranging from 0 (none) to 3 (high) with regard to the presence of epidermal, dermal, hypodermic and skin appendages atrophy as well as dermal and hypodermic sclerosis, according to Investigator's judgment.
Dermatology Life Quality Index (DLQI) | 6 months
  It is a simple 10-question validated questionnaire. The aim of the questionnaire is to measure how much patient's skin problem has affected patient's life. The scoring of each question is as follows:
  Very much scored 3 A lot scored 2 A little scored 1 Not at all scored 0 Not relevant scored 0 Question 7, 'prevented work or studying' scored 3 The DLQI is calculated by summing the score of each question resulting in a maximum of 30 and a minimumof 0. The higher the score, the more quality of life is impaired.
  HOW TO INTERPRET MEANING OF DLQI SCORES 0 - 1 no effect at all on patient's life 2 - 5 small effect on patient's life 6 - 10 moderate effect on patient's life 11 - 20 very large effect on patient's life 21 - 30 extremely large effect on patient's life

CONTACTS AND LOCATIONS:
Overall Officials: Simona Muratori, Dr, Principal Investigator — IRCCS Ca' Granda Osp. Maggiore Policlinico
Locations (1):
- IRCCS Ca' Granda Ospedale Maggiore Policlinico, Milan, Italy

IPD SHARING:
Plan to Share IPD: No